CLINICAL TRIAL: NCT06132828
Title: A Multicenter, Open-Label, Phase I Study to Evaluate the Safety, Tolerability, Pharmacokinetics of DR30206 in Patients With Advanced or Metastatic Solid Tumors
Brief Title: Evaluate the Safety, Tolerability, Pharmacokinetics of DR30206 in Patients With Advanced or Metastatic Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Zhejiang Doer Biologics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DR30206101
Record Dates: First submitted 2023-11-10; First posted 2023-11-15 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Solid Tumor
MeSH Terms: interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- DR30206 (Experimental): Subjects receive DR30206 monotherapy intravenously(IV) until no more benefits from treatment.
  Interventions: Drug: DR30206
- Phase Ib: DR30206 (Experimental): The non-small cell lung cancer subjects receive DR30206 (30mpk,Q3W) monotherapy intravenously(IV) until no more benefits from treatment.
  Interventions: Drug: DR30206

INTERVENTIONS:
Drug: DR30206 — Subjects receive DR30206 intravenously
  Other Names: DR30206 for Injection

SUMMARY:
This study is to characterize the safety,tolerability, pharmacokinetics(PK),and preliminary anti-tumor activity of DR30206, in subjects with advanced or metastatic solid tumors

DETAILED DESCRIPTION:
This study is an open, phase I study to evaluate the safety, tolerability, pharmacokinetics of DR30206 in patients with advanced or metastatic solid tumors. The study is composed of two parts: part A is Dose escalation stage and part B is Dose expansion stage

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign a written informed consent form
2. Patients must be ≥ 18 and ≤75 years of age
3. Part A: Subjects with advanced or metastatic malignant solid tumors confirmed by histology or cytology who have failed or are intolerant to standard therapy or have no effective standard therapy
4. Part B: The NSCLC cohort is planned to enroll patients with histologically or cytologically confirmed NSCLC who have locally advanced or metastatic NSCLC and are not eligible for curative treatment; patients must have no histologically confirmed EGFR-sensitive mutations or ALK gene fusions; they must not have received prior systemic anti-tumor therapy for locally advanced or metastatic NSCLC; and they must provide tumor tissue samples (approximately 5 unstained slides) obtained at the time of or after diagnosis of locally advanced or metastatic disease and within 2 years, without radiotherapy, which must be confirmed by the central laboratory to have tumor PD-L1 TPS ≥1%. Other potential cohorts may include patients with histologically or cytologically confirmed advanced or metastatic specific tumor types who have failed standard therapy, are intolerant to standard therapy, or have no effective standard therapy. These include, but are not limited to, cervical cancer, hepatocellular carcinoma, TNBC (Triple Negative Breast Cancer), and other tumor types such as gastric cancer, ovarian cancer, colorectal cancer, and tumor types with efficacy signals (CR/PR) identified during the dose escalation phase.
5. Patients in part A must have at least one evaluable lesion, and in part B must have at least one measurable lesion according to RECIST v1.1
6. Eastern Cooperative Oncology Group (ECOG) performance status (PS) score 0 or 1
7. The expected survival period ≥3 months
8. Adequate bone marrow, liver, and renal function
9. Male or female subjects with fertility must agree to take effective contraceptive measures during the study period and within 6 months after the end of the last medication
10. Be able to understand the procedures and methods of this study, and willing to strictly follow the clinical trial protocol to complete this study

Exclusion Criteria:

1. Patients with a history of severe allergies to monoclonal antibodies (mAb) or bispecific antibodies, or known allergies to drug component of the study drug
2. Patients with active malignant tumors within the past 2 years, except for the tumors participating in the study and locally cured tumors
3. Severe chronic or active infections, including but not limited to hospitalization due to complications of infection, bacteremia, or severe pneumonia, or any active infection that the investigator believes may affect the safety of the subject, within 4 weeks prior to the start of the study treatment; Systemic antibiotic treatment within 2 weeks before starting the study treatment
4. Received the following treatments or medications within 4 weeks before starting the study treatment: a. Interventional clinical studies; b. Major surgery or severe traumatic injury, or expected to require major surgery during the study process; c. Inoculate live attenuated vaccines, or expect to receive such vaccines during the study treatment period or within 5 months after the last administration of the study treatment; Systemic treatment with anti-tumor drugs, or local anti-tumor therapy, or treatment with systemic immune stimulators (including but not limited to interferon or interleukin-2 (IL-2)
5. Radical radiotherapy within 3 months before starting the study treatment
6. Received systemic immunosuppressive medication treatment within 4 weeks prior to the start of the study, or is expected to require systemic immunosuppressive medication during the study treatment period
7. Known active central nervous system (CNS) metastasis
8. There have been clinically significant cardiovascular and cerebrovascular diseases within 6 months prior to the first study drug dosing
9. Active stage of autoimmune disease or immune deficiency or history of autoimmune disease or immune deficiency
10. Have a history of interstitial pneumonia, idiopathic pulmonary fibrosis, organized pneumonia (such as bronchiolitis obliterans), drug-induced pneumonia, idiopathic pneumonia, or evidence of active pneumonia found on screening chest CT scans; Previously used hormone therapy for pneumonia
11. Active or previously diagnosed inflammatory bowel disease (such as Crohn's disease, ulcerative colitis)
12. During the screening period, there were a large or symptomatic moderate amount of pleural effusion, pericardial effusion, and abdominal effusion
13. During the screening period, imaging showed that the tumor were surrounded by important blood vessels or had obvious necrosis or cavities, and the investigators determined that enrolling into the study would pose a risk of bleeding
14. Previous or current complications such as gastrointestinal perforation surgery, wound healing, and bleeding events
15. Current or recent use of aspirin (>325 mg/day) or treatment with clopidogrel, clopidogrel, and cilostazol (within 10 days prior to the first study drug dosing)
16. Receiving full dose oral or parenteral anticoagulant or thrombolytic therapy, but still unstable for at least 2 weeks before the first study drug dosing
17. Adverse reactions caused by previous treatment that have not recovered to CTCAE 5.0 level 1 or below (but pigmentation, hair loss, etc. can be included if the investigator deems that there is no safety risk)
18. Known active infection
19. The subject has previously received allogeneic stem cell or organ transplantation
20. History of organ or hematopoietic stem cell transplantation that requires the use of immunosuppressants
21. Pregnant or lactating women, defined as women in a state of pregnancy until termination of pregnancy, are determined by laboratory human chorionic gonadotropin (hCG) testing within 7 days prior to the start of the study
22. Any other disease, medical condition or abnormality, metabolic dysfunction, alcohol or drug abuse or dependence, physical examination or lab testing results that potential impact on result interpretation or will increase the likelihood of complications for patients
23. Participants who are not appropriate for this clinical trial at the discretion of the investigator

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2023-11-27 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
PartA: Incidence of dose limiting toxicities (DLTs) | 21 days following first dose
  Dose-limiting describes side effects of a drug or other treatment that are serious enough to prevent an increase in dose or level of that treatment
PartA: Maximum tolerated dose (MTD) | 21 days following first dose
  As measured by number of participants experiencing dose related toxicity (DLT) in each escalating cohort
PartA: Recommend dose of expansion(RDE) | 21 days following first dose
  A Recommend dose of expansion will be determined based on safety data
PartA+B: Adverse evens (AEs) | Up to 90 days after last dose
  The incidence and severity of AEs graded according to NCI-CTCAE v5.0
PartA+B: Serious adverse evens (SAEs) | Up to 90 days after last dose
  A Serious Adverse Event (SAE) is an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect
PartB: Objective response rate (ORR) | Up to approximately 12 months
  Objective response rate (ORR) is the proportion of subjects with complete response (CR) or partial response (PR), based on RECIST v1.1
PartB: Recommended phase 2 dose (RP2D) | 21 days following first dose
  A recommended phase 2 dose will be determined based on safety data

CONTACTS AND LOCATIONS:
Overall Officials: Caicun Zhou, MD, Principal Investigator — Shanghai Pulmonary Hospital, Shanghai, China; Yanshan Huang, PhD, Study Chair — Zhejiang Doer Biologics Co., Ltd.; Junfang Xu, MD, Study Director — Huadong Medicine Co., Ltd.
Locations (1):
- Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No